CLINICAL TRIAL: NCT01200693
Title: Z-SEA-SIDE: Sirolimus Versus Everolimus Versus Zotarolimus-eluting Stent Assessment in Bifurcated Lesions and Clinical SIgnificance of Residual siDE-branch Stenosis
Acronym: Z-SEA-SIDE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Francesco Burzotta, MD, PhD, Catholic University of the Sacred Heart
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSC-002
Record Dates: First submitted 2010-06-10; First posted 2010-09-14 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Coronary Artery Disease; Coronary Stenosis
Keywords: Angioplasty, Transluminal, Percutaneous Coronary; Drug-Eluting Stents
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ZES (Active Comparator): Patients with coronary bifurcation lesions treated by Zotarolimus eluting stent
  Interventions: Device: Zotarolimus eluting stent
- SES (Active Comparator): Patients with coronary bifurcation lesions treated by Sirolimus eluting stent
  Interventions: Device: Sirolimus eluting stent
- EES (Active Comparator): Patients with coronary bifurcation lesions treated by Everolimus eluting stent
  Interventions: Device: Everolimus eluting stent

INTERVENTIONS:
Device: Sirolimus eluting stent — Implantation of Sirolimus eluting stent
  Other Names: Cypher stent - Cordis (Johnson&Johnson Company)
  Arms: SES
Device: Everolimus eluting stent — Implantation of Everolimus eluting stent
  Other Names: Xience stent - Abbot company
  Arms: EES
Device: Zotarolimus eluting stent — Implantation of Zotarolimus eluting stent
  Other Names: Endeavor Resolute stent - Medtronic company
  Arms: ZES

SUMMARY:
BACKGROUND:

Bifurcated lesions are a challenging subset in percutaneous coronary interventions (PCI). The selection of the type of drug-eluting stents (DES) and the technique for stent implantation have not been clarified. The side-branch (SB) is emerging as critical point, accounting for more than a third of the significant restenosis in the DES era. A series of data supports the adoption of a conservative strategy: stenting the main vessel (MV) only and reserving a conservative approach on the SB. Yet, the clinical relevance in terms of inducible ischemia of sub-optimal angiographic result has not been clarified.

AIMS OF THE STUDY:

The aims of the present study are:

1. to compare in a prospective study the acute 3D angiographic results and the late clinical outcome of Sirolimus-eluting (SES) vs Everolimus-eluting (EES) vs Zotarolimus eluting stent (ZES) obtained using a provisional TAP-stenting technique.
2. to prospectively assess the clinical relevance (inducible ischemia) of suboptimal angiographic result in the SB after stenting.

METHODS TO BE APPLIED:

75 consecutive patients with bifurcated lesions undergoing PCI with the provisional T-and-small-protruding (TAP) technique with ZES implantation will be enrolled. Procedural and post-PCI details will be prospectively recorded. The subgroup of patients in which complete revascularization has been achieved will enter a systematic assessment of inducible ischemia by early and late exercise tests.

Off line 3D quantitative coronary angiography (QCA) assessment will be performed and used to divide the study population in 2 groups according to the SB residual stenosis:

* Group O (optimal SB angiographic result): post-PCI SB area stenosis<50%
* Group S (sub-optimal SB angiographic result): post-PCI SB area stenosis>50%.

For the comparison among SES and EES, data will be obtained from the randomized trial SEA-SIDE (NCT00697372).

PRIMARY STUDY END-POINTS.

1. COMPARISON BETWEEN ZES, SES AND EES:

   SB acute angiographic result; SB trouble; target bifurcation failure.
2. SB-RELATED ISCHAEMIA of Group O vs Group S in patients with complete revascularization: inducible ischemia at the early exercise test or occurrence of early spontaneous ischemia related to the SB.

DETAILED DESCRIPTION:
Bifurcated lesions are challenging target lesions in percutaneous coronary interventions (PCI) which may specifically benefit from the usage of drug-eluting stents (DES). However, the selection of the type of DES and the technique for DES implantation have not been clarified. In spite of the technique adopted, the side-branch (SB) is emerging as critical point, accounting for more than a third of the significant restenosis in the DES era. A series of data supports the adoption of a conservative strategy: stenting the main vessel (MV) only and reserving a conservative approach on the SB as this is not associated with worse outcome compared to more complex stenting strategies. Yet, the clinical relevance in terms of inducible ischemia of sub-optimal angiographic result has not been clarified.

AIMS OF THE STUDY:

The aims of the present study are:

1. to compare in a prospective study the acute 3D angiographic results (as a measure of the impact of stent design) and the late clinical outcome of Sirolimus-eluting (SES) vs Everolimus-eluting (EES) vs Zotarolimus-eluting stent (ZES) obtained using a provisional T-and-small-protruding (TAP) approach to treat bifurcated lesions.
2. to prospectively assess the clinical relevance (in terms of inducible ischemia) of suboptimal angiographic result in the SB of bifurcated lesions treated by stenting.

METHODS TO BE APPLIED:

75 consecutive patients with bifurcated lesions undergoing PCI with the provisional TAP-stenting technique with ZES implantation will be enrolled. Procedural details, post-PCI cardiac enzyme release, clinical outcome up to 1 year will be prospectively recorded. After the procedure, the subgroup of patients in which complete revascularization has been achieved (no untreated stenosis >50% in any other vessel, no residual stenosis >50% in any other treated vessel), will enter a systematic assessment of inducible ischemia by early (<8 days) and late (6-month) exercise tests.

Off line 3D quantitative coronary angiography (QCA) assessment will be performed and used to divide the study population in 2 groups according to the SB residual stenosis: Group O (optimal SB angiographic result): post-PCI SB area stenosis<50% and Group S (sub-optimal SB angiographic result): post-PCI SB area stenosis>50%.

For the comparison among SES and EES, data will be obtained from the randomized trial SEA-SIDE (NCT00697372).

PRIMARY STUDY END-POINTS.

1.

COMPARISON BETWEEN ZES, SES AND EES:

* "SB acute angiographic result": comparison of the 3DQCA-estimated MLD and MLA in the SB.
* "SB trouble": composite of: 1. occurrence of SB TIMI flow <3 after MV stenting throughout the procedure; 2. need of guidewire(s) different from BMW to re-wire SB after MV stenting; 3. failure to re-wire the SB after MV stenting; 4. failure to dilate the SB after MV stenting and SB re-wiring.
* target bifurcation failure (TBF) defined as target bifurcation-related major adverse coronary events (MACE) or target bifurcation angiographic failure.

  2. SB-RELATED ISCHAEMIA of Group O vs Group S in patients with complete revascularization: inducible ischemia (diagnostic ST-segment changes) at the early (<8 days) exercise test or occurrence of early (<12 weeks) spontaneous ischemia related to the SB (any ischemic episode requiring unplanned coronary angiography with documentation of main vessel patency).

ELIGIBILITY:
Inclusion Criteria:

* de novo bifurcated lesions
* lesions >50% located in a major bifurcation point
* TIMI >2 on both main vessel and side branch
* main vessel visual diameter >2.5 mm
* side branch visual diameter >2.0 mm
* >18 years of age
* signed the informed consent to enter the study

Exclusion Criteria:

* known hypersensitivity to Sirolimus, Everolimus, cobalt, chromium, nickel, tungsten acrylic and fluoro-polymers
* contraindications to double antiplatelet therapy acute (within 48 hours) ST-elevation acute myocardial infarction

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-11; Primary Completion 2010-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
6-9-12-18 MONTH CLINICAL OUTCOME | 18 MONTHS
ACUTE ANGIOGRAPHIC RESULT | 7 DAYS
  * "MV acute angiographic result": comparison of the 3DQCA-estimated MLD and MLA in the MV.
  * "SB acute angiographic result": comparison of the 3DQCA-estimated MLD and MLA in the SB.
SIDE BRANCH TROUBLE | 7 DAYS
  "SB trouble" composite of:
  1. occurrence of SB TIMI flow <3 after MV stenting throughout the procedure;
  2. need of guidewire(s) different from BMW to re-wire SB after MV stenting;
  3. failure to re-wire the SB after MV stenting;
  4. failure to dilate the SB after MV stenting and SB re-wiring.
TARGET BIFURCATION FAILURE | 18 MONTHS
  - target bifurcation failure (TBF) defined as target bifurcation-related major adverse coronary events (MACE) or target bifurcation angiographic failure.

SECONDARY OUTCOMES:
TECHNICAL CHARACTERISTICS | 7 DAYS
  comparison of procedural time, fluoroscopy time, total x-ray exposure, contrast media volume usage, number of guidewires used to wire the SB, direct stenting failure rate, kissing balloon rate, occurrence of transient deterioration of blood flow through the SB (TIMI<3)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Burzotta, MD,PhD,FESC, Principal Investigator — Catholic University of Sacred Heart
Locations (1):
- Institute of Cardiology - Catholic University of Sacred Heart, Rome, Italy

REFERENCES:
- [Background] Colombo A, Moses JW, Morice MC, Ludwig J, Holmes DR Jr, Spanos V, Louvard Y, Desmedt B, Di Mario C, Leon MB. Randomized study to evaluate sirolimus-eluting stents implanted at coronary bifurcation lesions. Circulation. 2004 Mar 16;109(10):1244-9. doi: 10.1161/01.CIR.0000118474.71662.E3. Epub 2004 Feb 23. PMID 14981005
- [Background] Ormiston JA, Webster MW, El Jack S, Ruygrok PN, Stewart JT, Scott D, Currie E, Panther MJ, Shaw B, O'Shaughnessy B. Drug-eluting stents for coronary bifurcations: bench testing of provisional side-branch strategies. Catheter Cardiovasc Interv. 2006 Jan;67(1):49-55. doi: 10.1002/ccd.20453. PMID 16003787
- [Background] Pan M, Suarez de Lezo J, Medina A, Romero M, Delgado A, Segura J, Ojeda S, Mazuelos F, Hernandez E, Melian F, Pavlovic D, Esteban F, Herrador J. Drug-eluting stents for the treatment of bifurcation lesions: a randomized comparison between paclitaxel and sirolimus stents. Am Heart J. 2007 Jan;153(1):15.e1-7. doi: 10.1016/j.ahj.2006.10.017. PMID 17174630
- [Background] Lefevre T, Louvard Y, Morice MC, Loubeyre C, Piechaud JF, Dumas P. Stenting of bifurcation lesions: a rational approach. J Interv Cardiol. 2001 Dec;14(6):573-85. doi: 10.1111/j.1540-8183.2001.tb00375.x. PMID 12053378
- [Background] Ge L, Tsagalou E, Iakovou I, Sangiorgi GM, Corvaja N, Airoldi F, Chieffo A, Montorfano M, Michev I, Colombo A. In-hospital and nine-month outcome of treatment of coronary bifurcational lesions with sirolimus-eluting stent. Am J Cardiol. 2005 Mar 15;95(6):757-60. doi: 10.1016/j.amjcard.2004.11.030. PMID 15757605
- [Background] Valgimigli M, Malagutti P, Rodriguez Granillo GA, Tsuchida K, Garcia-Garcia HM, van Mieghem CA, Van der Giessen WJ, De Feyter P, de Jaegere P, Van Domburg RT, Serruys PW. Single-vessel versus bifurcation stenting for the treatment of distal left main coronary artery disease in the drug-eluting stenting era. Clinical and angiographic insights into the Rapamycin-Eluting Stent Evaluated at Rotterdam Cardiology Hospital (RESEARCH) and Taxus-Stent Evaluated at Rotterdam Cardiology Hospital (T-SEARCH) registries. Am Heart J. 2006 Nov;152(5):896-902. doi: 10.1016/j.ahj.2006.03.029. PMID 17070153
- [Background] Iakovou I, Ge L, Colombo A. Contemporary stent treatment of coronary bifurcations. J Am Coll Cardiol. 2005 Oct 18;46(8):1446-55. doi: 10.1016/j.jacc.2005.05.080. Epub 2005 Sep 28. PMID 16226167
- [Background] Pan M, de Lezo JS, Medina A, Romero M, Segura J, Pavlovic D, Delgado A, Ojeda S, Melian F, Herrador J, Urena I, Burgos L. Rapamycin-eluting stents for the treatment of bifurcated coronary lesions: a randomized comparison of a simple versus complex strategy. Am Heart J. 2004 Nov;148(5):857-64. doi: 10.1016/j.ahj.2004.05.029. PMID 15523318
- [Background] Ge L, Iakovou I, Cosgrave J, Agostoni P, Airoldi F, Sangiorgi GM, Michev I, Chieffo A, Montorfano M, Carlino M, Corvaja N, Colombo A. Treatment of bifurcation lesions with two stents: one year angiographic and clinical follow up of crush versus T stenting. Heart. 2006 Mar;92(3):371-6. doi: 10.1136/hrt.2005.061531. Epub 2005 Jun 17. PMID 15964941
- [Background] Steigen TK, Maeng M, Wiseth R, Erglis A, Kumsars I, Narbute I, Gunnes P, Mannsverk J, Meyerdierks O, Rotevatn S, Niemela M, Kervinen K, Jensen JS, Galloe A, Nikus K, Vikman S, Ravkilde J, James S, Aaroe J, Ylitalo A, Helqvist S, Sjogren I, Thayssen P, Virtanen K, Puhakka M, Airaksinen J, Lassen JF, Thuesen L; Nordic PCI Study Group. Randomized study on simple versus complex stenting of coronary artery bifurcation lesions: the Nordic bifurcation study. Circulation. 2006 Oct 31;114(18):1955-61. doi: 10.1161/CIRCULATIONAHA.106.664920. Epub 2006 Oct 23. PMID 17060387
- [Background] Koo BK, Kang HJ, Youn TJ, Chae IH, Choi DJ, Kim HS, Sohn DW, Oh BH, Lee MM, Park YB, Choi YS, Tahk SJ. Physiologic assessment of jailed side branch lesions using fractional flow reserve. J Am Coll Cardiol. 2005 Aug 16;46(4):633-7. doi: 10.1016/j.jacc.2005.04.054. PMID 16098427
- [Background] Burzotta F, Gwon HC, Hahn JY, Romagnoli E, Choi JH, Trani C, Colombo A. Modified T-stenting with intentional protrusion of the side-branch stent within the main vessel stent to ensure ostial coverage and facilitate final kissing balloon: the T-stenting and small protrusion technique (TAP-stenting). Report of bench testing and first clinical Italian-Korean two-centre experience. Catheter Cardiovasc Interv. 2007 Jul 1;70(1):75-82. doi: 10.1002/ccd.21194. PMID 17585382
- [Background] Gradaus R, Mathies K, Breithardt G, Bocker D. Clinical assessment of a new real time 3D quantitative coronary angiography system: evaluation in stented vessel segments. Catheter Cardiovasc Interv. 2006 Jul;68(1):44-9. doi: 10.1002/ccd.20775. PMID 16770813
- [Derived] Burzotta F, Trani C, Talarico GP, Tommasino A, Todaro D, Coluccia V, Pirozzolo G, Niccoli G, Leone AM, Porto I, Schiavoni G, Crea F. Resolute zotarolimus-eluting stent to treat bifurcated lesions according to the provisional technique: a procedural performance comparison with sirolimus- and everolimus-eluting stents. Cardiovasc Revasc Med. 2013 May-Jun;14(3):122-7. doi: 10.1016/j.carrev.2013.01.002. Epub 2013 Feb 27. PMID 23453789